CLINICAL TRIAL: NCT04502368
Title: Fiberoptic Bronchoscopy and Bronchoalveolar Lavage in Critically Ill Ventilated Patients: Impact on Respiratory Mechanics and Gas Exchange
Brief Title: Fiberoptic Bronchoscopy and Bronchoalveolar Lavage in Critically Ill Ventilated Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Erasme University Hospital (Other)
Responsible Party: Principal Investigator, Francesco Ricottilli, MD, Resident, Erasme University Hospital
Other Study IDs: SRB2020-289; P2020/375 (Other: Erasme - ULB Ethics Committee)
Record Dates: First submitted 2020-08-03; First posted 2020-08-06 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Fiberoptic Bronchoscopy (FOB); Bronchoalveolar Lavage (BAL); Respiratory Disease
Keywords: Respiratory Insufficiency; Respiratory Distress Syndrome; Mechanical Ventilation; COVID-19; Fiberoptic Bronchoscopy (FOB); Bronchoalveolar Lavage (BAL)
MeSH Terms: conditions — Respiration Disorders; Respiratory Insufficiency; Respiratory Distress Syndrome; COVID-19 | interventions — Bronchoalveolar Lavage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Fiberoptic Bronchoscopy (FOB) — FOB under full sedation (RASS sedation scale -5) and full paralysis.
Procedure: Bronchoalveolar Lavage (BAL) — BAL under full sedation (RASS sedation scale -5) and full paralysis. Lavage: NaCl 0,9% 50ml x 3 in lung region targetted according to RX/CT scan.
Diagnostic Test: Electrical Impedance Tomography (EIT) — Realtime thoracic impedance coupled with ventilation parameters recording.
  Other Names: PulmoVista® 500 - Draeger
Diagnostic Test: Arterial Blood Gas test (ABG) — Multiples Arterial Blood Gas test (ABG) via arterial catheter.

SUMMARY:
Fiberoptic bronchoscopy (FOB) is widely used as a diagnostic or therapeutic procedure in intensive care units. Patients with ARDS or COVID-19 disease often undergoes to these procedures. However, intensive care patients might suffer from serious side effects such as prolonged oxygen desaturation and adverse change in lung compliance and resistance. This study aims to evaluate these changes and determine their impact on patient stability.

DETAILED DESCRIPTION:
Fiberoptic bronchoscopy (FOB) is widely used in intensive care units as a diagnostic or therapeutic procedure. FOB in respiratory failure patients supported by mechanical ventilation may worsen hypoxemia and hypercapnia, therefore FOB requires careful consideration in this patient population. The generally accepted indications for FOB in ventilated patients are removal of retained secretions, resolution of atelectasis and evaluation of hemoptysis. A diagnostic indication is the bronchoalveolar lavage (BAL), to sample the lower respiratory tract without contamination. Studies of FOB performed in mechanically ventilated patients suggest an acceptable safety profile, except for the occurrence of hypoxemia as the main adverse event. Bronchoalveolar Lavage (BAL) in normal volunteers is reported to be safe and does not lead to measurable changes in pulmonary function parameters. However, in intensive care patients may suffer from serious side effects such as prolonged oxygen desaturation. Moreover, reductions in arterial oxygen tension (PaO2) have been reported to persist in some patients for 4 h and more after the procedure. Authors reported the BAL procedure is associated to a worsening of PaO2/FiO2 ratio, in several ARDS patients the drop in PaO2 was higher than 30%. Moreover a physiological study in patients undergoing FOB and BAL showed adverse change in lung compliance and resistance.

The purpose of this prospective study is to determine the alterations in respiratory mechanics (regional compliance and resistance) and gas exchange induced by FOB and BAL up to 6 hours after the procedure. The lung regional ventilation evaluation will be made by electrical impedance tomography (EIT).

ELIGIBILITY:
Inclusion Criteria:

Mechanically ventilated ICU patients requiring a FOB or FOB + BAL

Exclusion Criteria:

* PaO2/FiO2 ratio <100
* Age < 18 years
* Pregnancy
* Unstable angina and recent (less than 1 week) myocardial infarction
* Uncontrolled cranial hypertension
* Major hemodynamic instability
* Any previous lung surgery (except for lung transplantation)
* Obesity (BMI > 50)
* Chest circumference > 150 cm
* Electronic implanted device (pacemaker, neurostimulator, etc.)

Patients who had undergone several bronchoscopy procedures could not be included twice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intensive Care Unit admitted patients
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-03-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Regional Compliance Variation | From FOB/BAL to 6 hours later
  The variation of regional compliance, calculated by electrical impedance

SECONDARY OUTCOMES:
Regional Resistance Variation | From FOB/BAL to 6 hours later
  The variation of regional resistance, calculated by electrical impedance
Regional Compliance and FOB duration | From FOB/BAL to 6 hours later
  Relation between regional compliance variation and FOB duration
Regional Compliance and PaO2 | From FOB/BAL to 6 hours later
  Relation between regional compliance variation and PaO2 variation
Atelectasis areas and BAL flooded areas | From FOB/BAL to 6 hours later
  Relation between atelectasis impedance-detected areas and BAL flooded impedance-detected areas
PaO2 and PaO2/FiO2 ratio | From FOB/BAL to 6 hours later
  Variation of PaO2 and PaO2/FiO2 ratio post FOB/BAL
PaCO2 | From FOB/BAL to 6 hours later
  Variation of PaCO2 post FOB/BAL
Endotracheal tube size and Fiberscope size | From FOB/BAL to 6 hours later
  Relation between the endotracheal tube/fiberscope size ratio and gas exchanges
Hemodynamic variations | From FOB/BAL to 6 hours later
  Heart rate (HR), Blood Pressure (BP)

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Ricottilli, MD, Principal Investigator — Intensive Care Unit - Erasme University Hospital; Leda Nobile, MD, Principal Investigator — Intensive Care Unit - Erasme University Hospital
Locations (1):
- Erasme University Hospital - Intensive Care Unit, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Du Rand IA, Blaikley J, Booton R, Chaudhuri N, Gupta V, Khalid S, Mandal S, Martin J, Mills J, Navani N, Rahman NM, Wrightson JM, Munavvar M; British Thoracic Society Bronchoscopy Guideline Group. British Thoracic Society guideline for diagnostic flexible bronchoscopy in adults: accredited by NICE. Thorax. 2013 Aug;68 Suppl 1:i1-i44. doi: 10.1136/thoraxjnl-2013-203618. No abstract available. PMID 23860341
- [Background] Kamel T, Helms J, Janssen-Langenstein R, Kouatchet A, Guillon A, Bourenne J, Contou D, Guervilly C, Coudroy R, Hoppe MA, Lascarrou JB, Quenot JP, Colin G, Meng P, Roustan J, Cracco C, Nay MA, Boulain T; Clinical Research in Intensive Care Sepsis Group (CRICS-TRIGGERSEP). Benefit-to-risk balance of bronchoalveolar lavage in the critically ill. A prospective, multicenter cohort study. Intensive Care Med. 2020 Mar;46(3):463-474. doi: 10.1007/s00134-019-05896-4. Epub 2020 Jan 7. PMID 31912201
- [Background] Bauer TT, Torres A, Ewig S, Hernandez C, Sanchez-Nieto JM, Xaubet A, Agusti C, Rodriguez-Roisin R. Effects of bronchoalveolar lavage volume on arterial oxygenation in mechanically ventilated patients with pneumonia. Intensive Care Med. 2001 Feb;27(2):384-93. doi: 10.1007/s001340000781. PMID 11396283
- [Background] Trouillet JL, Guiguet M, Gibert C, Fagon JY, Dreyfuss D, Blanchet F, Chastre J. Fiberoptic bronchoscopy in ventilated patients. Evaluation of cardiopulmonary risk under midazolam sedation. Chest. 1990 Apr;97(4):927-33. doi: 10.1378/chest.97.4.927. PMID 2108848
- [Background] Klein U, Karzai W, Zimmermann P, Hannemann U, Koschel U, Brunner JX, Remde H. Changes in pulmonary mechanics after fiberoptic bronchoalveolar lavage in mechanically ventilated patients. Intensive Care Med. 1998 Dec;24(12):1289-93. doi: 10.1007/s001340050764. PMID 9885882
- [Background] Costa EL, Borges JB, Melo A, Suarez-Sipmann F, Toufen C Jr, Bohm SH, Amato MB. Bedside estimation of recruitable alveolar collapse and hyperdistension by electrical impedance tomography. Intensive Care Med. 2009 Jun;35(6):1132-7. doi: 10.1007/s00134-009-1447-y. Epub 2009 Mar 3. PMID 19255741